CLINICAL TRIAL: NCT04400253
Title: A Multilevel Physical Activity Intervention for South Asian Women and Girls (SAATH)
Brief Title: South Asians Active Together (SAATH) Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern University (Other)
Collaborators: Skokie Health Department (Unknown); Skokie Park District (Unknown); University of Illinois at Chicago (Other); Metropolitan Asian Family Services (Unknown); University of Chicago (Other); Ann & Robert H Lurie Children's Hospital of Chicago (Other)
Responsible Party: Principal Investigator, Namratha Kandula, Prinicipal Investigator, Northwestern University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: STU00211374:
Record Dates: First submitted 2020-05-11; First posted 2020-05-22 (Actual); Last update posted 2024-11-22 (Actual); Status verified 2024-11

CONDITIONS: Physical Inactivity; South Asian
MeSH Terms: conditions — Sedentary Behavior

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): The intervention group will receive a 18-week in-person program. The program includes the following components: multi family group counseling, group exercise classes, mother group discussion, daughter group discussion and Fitbit.
  Interventions: Behavioral: SAATH Intervention
- Control group (No Intervention): The group group will receive print materials about physical activity.

INTERVENTIONS:
Behavioral: SAATH Intervention — SAATH intervention is a physical activity intervention for South Asian mothers and daughters with group exercise classes and discussion groups.
  Arms: Intervention group

SUMMARY:
South Asian immigrant women and girls are at increased risk for insufficient physical activity and are not being reached by current approaches to physical activity promotion. This randomized control trial study will test the effectiveness and implementation of a multi component physical activity intervention directed at the environment, family, interpersonal and individual levels to promote physical activity among South Asian immigrant mothers and daughters.

ELIGIBILITY:
The sample of this study is South Asian mothers and their daughters. The inclusion criteria for the mother include:

* Identifying herself as South Asian,
* having a sedentary lifestyle as assessed using a self-report questionnaire
* having ability to communicate in Hindi, Gujarati, Urdu, or English.
* Having a daughter aged 11-16 years

Exclusion Criteria:

* having known medical condition that restricts ability to participate in moderate intensity Physical Activity
* Unable to complete study procedures (including not wearing accelerometer during run-in)
* Currently pregnant
* Unable to provide informed consent or assent.

Min Age: 11 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — South Asian girls and women
Enrollment: 252 (Actual)
Dates: Start 2020-08-01 (Actual); Primary Completion 2024-03-26 (Actual); Study Completion 2024-03-26 (Actual)

PRIMARY OUTCOMES:
Averaged daily minutes spent in moderate- and vigorous-intensity physical activity measured by ActiGraph accelerometers | The outcome will be assessed before the intervention (week 0) and after the intervention (week 18)
  Moderate- and vigorous-intensity physical activity will be identified based on the accelerometer count cut-point for moderate intensity and daily minutes spent in moderate- and vigorous-intensity physical activity estimated for seven days will be averaged

SECONDARY OUTCOMES:
Averaged daily minutes spent in walking or running behavior measured by ActiGraph accelerometers | The outcome will be assessed before the intervention (week 0) and after the intervention (week 18)
  Walking and running behavior will be recognized using a machine learning activity recognition algorithm and daily minutes spent in walking or running behavior estimated for seven days will be averaged
Averaged daily hours spent in sedentary behaviors measured by ActiGraph accelerometers | The outcome will be assessed before the intervention (week 0) and after the intervention (week 18)
  Sedentary behaviors will be identified based on the accelerometer count cut-point for sedentary behaviors and daily minutes spent in sedentary behaviors estimated for seven days will be averaged
Systolic and diastolic blood pressure (mmHg) measured by a sphygmomanometer | The outcome will be assessed before the intervention (week 0) and after the intervention (week 18)
  Blood pressure will be measured three times while sitting down and relaxing on a chair and the last two measures will be averaged
Self-efficacy score measured by the Exercise Confidence Survey | The outcome will be assessed before the intervention (week 0) and after the intervention (week 18)
  The self-efficacy score will be calculated by averaging the responses (scored 1 to 5 point for the responses of strongly disagree to strongly agree) from each question item
Self-efficacy score measured by Dishman's Barriers to Self-Efficacy questionnaire | The outcome will be assessed before the intervention (week 0) and after the intervention (week 18)
  The self-efficacy score will be calculated by averaging the responses (scored 1 to 5 point; higher scores mean higher self-efficacy [a better outcome])

CONTACTS AND LOCATIONS:
Overall Officials: Namratha Kandula, MD, MPH, Principal Investigator — Northwestern University
Locations (1):
- Northwestern University-Feinberg School of Medicine, Chicago, Illinois, United States